CLINICAL TRIAL: NCT05172154
Title: GlowTest COVID-19 Antigen Home Test Kit Usability
Brief Title: GlowTest COVID-19 Antigen Home Test Kit Usability Study
Status: Completed | Type: Observational
Sponsor: Arion Bio (Industry)
Collaborators: CSSi Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-001-02
Record Dates: First submitted 2021-12-24; First posted 2021-12-29 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 15 subjects testing themselves: 15 subjects 14 years of age and older
  Interventions: Diagnostic Test: GlowTest COVID-19 Antigen Home Test Kit
- 15 subjects testing someone else: 15 adult subjects testing individuals ages 2-13
  Interventions: Diagnostic Test: GlowTest COVID-19 Antigen Home Test Kit

INTERVENTIONS:
Diagnostic Test: GlowTest COVID-19 Antigen Home Test Kit — The Arion Bio GlowTest COVID-19 Antigen Home Test is a lateral flow immunoassay intended for the qualitative detection of SARS-CoV-2 nucleocapsid protein antigens from individuals with or without symptoms or other epidemiological reasons to suspect a COVID-19 infection

SUMMARY:
The purpose of this study is to evaluate the usability of the GlowTest COVID-19 Antigen Home Test in Home Use.

DETAILED DESCRIPTION:
The Arion Bio GlowTest COVID-19 Antigen Home Test is a lateral flow immunoassay intended for the qualitative detection of SARS-CoV-2 nucleocapsid protein antigens from individuals with or without symptoms or other epidemiological reasons to suspect a COVID-19 infection. The test is intended for non-prescription home use with self collected direct anterior nares swab samples from individuals ages 14 years and older or adult collected anterior nares swab samples from individuals aged 2 to 13.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent/assent is signed and dated prior to any study-related activities.
2. Male and female Subjects 2 years of age and older.
3. Subject is willing to provide a self-collected nasal swab sample. (If under the age of 14, the sample will be collected by an adult.)
4. Subject agrees to complete all aspects of the study.

Exclusion Criteria:

1. Subject has a visual impairment that cannot be restored with glasses or contact lenses.
2. Subject has prior medical or laboratory training.
3. Subject uses home diagnostics, e.g., glucose meters, HIV tests.
4. Subject has prior experience with home COVID test kits

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A minimum of 30 completed subjects with a minimum of 15 subjects testing themselves and a minimum of 15 subjects testing another person (child).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Assess the usability of the Quick Reference Instructions (QRI) based upon observer evaluation. | 90 minutes
  Track the percentage of subjects who perform the test correctly and according to the QRI.
Assess the usability of the kit for home use based upon participant evaluation | 90 minutes
  Track usability of the test by asking subjects a series of questions regarding the ease of use of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Geller, MD, Principal Investigator — Centennial Medical Group
Locations (1):
- Centennial Medical, Elkridge, Maryland, United States

IPD SHARING:
Plan to Share IPD: No